CLINICAL TRIAL: NCT01750489
Title: Skeletal and Respiratory Muscle Dysfunction in Patients With COPD: the Role of Sympathetic Activation
Brief Title: Muscle Dysfunction in Patients With Chronic Obstructive Lung Disease (COPD): the Role of Sympathetic Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Tobias Raupach, Dr., University Medical Center Goettingen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA1937/1-1
Record Dates: First submitted 2012-12-09; First posted 2012-12-17 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- COPD (No Intervention)
- COPD with non-invasive ventilation (NIV) (Experimental): Starting non-invasive ventilation with the patient's own device during registration of MSNA.
  Interventions: Device: non-invasive ventilation (NIV)
- Healthy control subjects (No Intervention)

INTERVENTIONS:
Device: non-invasive ventilation (NIV)
  Arms: COPD with non-invasive ventilation (NIV)

SUMMARY:
The objective of the project is to better understand the causes of exercise limitation, dyspnea and neurohumoral activation in patients with COPD. In particular, the investigators aim to explore the mutual interaction of neurohumoral activation and exercise limitation thereby focussing on differential effects of the peripheral muscle and the diaphragm.

Eventually the findings might influence treatment modalities. If sympathetic activation contributes to exercise limitation then drugs influencing the autonomic nervous system would be a reasonable therapeutic concept. If a reduction of sympathetic activity due to an alteration of the ergoreflex can be achieved by non-invasive ventilation this would help to improve dyspnea and exercise capacity.

DETAILED DESCRIPTION:
Our aim is to investigate whether reduced exercise capacity, increased respiratory drive and dyspnoea are linked to heightened sympathetic activation at rest and during exercise in patients with COPD. Furthermore, the effect of unloading the respiratory muscles by using non-invasive ventilation (NIV) will be assessed. Fifteen stable COPD patients without NIV will be matched to 15 healthy control subjects (with sufficient microneurography recording). Furthermore COPD patients on regular NIV will be studied. Each participant will undergo symptom limited bicycle exercise and a handgrip protocol. Microneurography will be used to quantify sympathetic activity by the transcutaneous registration of postganglionic sympathetic efferents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD II or III according to the GOLD guidelines
* FEV1 of less than 60% of the predicted value
* RV/TLC > 45%
* Optimal stable medication according to the GOLD guidelines for at least 2 weeks
* The last exacerbation must not be more recent than three weeks
* Stable sinus rhythm
* The subgroup on NIV should be stable on NIV for > 1 month

Exclusion Criteria:

* not willing or unable to sign the informed consent before the study begins
* Age under 30 or over 80 years
* paO2< 55 mmHg or PaCO2 > 45 mmHg on arterial blood gas analysis (For patients on NIV, PaCO2 values of up to 55 mmHg are acceptable.)
* Treatment with drugs having direct sympathomimetic activity (e.g. theophylline, moxonidine, clonidine)
* Oral medication with beta2 sympathomimetics (therapy with long-acting inhaled beta2 sympathomimetics is permitted)
* History of sleep apnoea or documented evidence of > 15 episodes of apneas and/or hypopnea per hour during sleep. An episode of apnea is defined as the cessation of inspiratory airflow for 10 s or more. Hypopnea is defined as a reduction in airflow (> 50%) lasting for more than 10 s in comparison with the maximum airflow recorded during the preceding breathing cycle.
* Myocardial infarction (MI) or a coronary revascularization procedure within the previous 2 calendar months
* Clinically evident polyneuropathy
* Diabetes mellitus necessitating any pharmacologic therapy
* Severe (i.e., life-limiting) concomitant disease, including life-threatening malignancy (cancer likely to reduce life expectancy to less than 5 years), acquired immune deficiency syndrome, or any other life-threatening disease.
* Diuretics should not be taken before measurements

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2011-08; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
muscle sympathetic nerve activity (MSNA) | 90 minutes
  In a 90 minute microneurographic measurement muscle sympathetic nerve activity is assessed.
Arterial stiffness | 90 min

SECONDARY OUTCOMES:
VE/VCO2 | During 8-15 minutes bicycle exercise

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Andreas, Professor, Principal Investigator — Universitaetsmedizin Goettingen
Locations (1):
- Universitaetsmedizin Goettingen, Göttingen, Germany

REFERENCES:
- [Background] Raupach T, Bahr F, Herrmann P, Luethje L, Heusser K, Hasenfuss G, Bernardi L, Andreas S. Slow breathing reduces sympathoexcitation in COPD. Eur Respir J. 2008 Aug;32(2):387-92. doi: 10.1183/09031936.00109607. Epub 2008 Apr 2. PMID 18385175
- See also: Information about research facility — http://www.lungenfachklinik-immenhausen.de/
- See also: Information about research facility — http://www.med.uni-goettingen.de